CLINICAL TRIAL: NCT00628862
Title: A 12-week, Randomised, Double-blind, Placebo-controlled, Parallel-group, Multi-national, Phase III, Efficacy and Safety Study of Inhaled Formoterol 4.5 μg and 9 μg Twice Daily in Japanese and European Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Evaluation of Efficacy and Safety of Formoterol in Patients With COPD Compared With Placebo in Patients in Japan, EU
Acronym: OCEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5122C00001; EudraCT no 2007-003999-19
Record Dates: First submitted 2008-01-24; First posted 2008-03-05 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- F 4.5 bid (Experimental): Formoterol 4.5 ug twice daily (bid)
  Interventions: Drug: Formoterol Turbuhaler® 4.5mg
- F 9.0 bid (Experimental): Formoterol 9.0 ug bid
  Interventions: Drug: Formoterol Turbuhaler® 9 mg
- PBO (Placebo Comparator): Placebo
  Interventions: Drug: Turbuhaler® placebo

INTERVENTIONS:
Drug: Formoterol Turbuhaler® 4.5mg — 4.5 mg inhaled twice daily
  Other Names: Oxis
  Arms: F 4.5 bid
Drug: Formoterol Turbuhaler® 9 mg — 9 mg inhaled twice daily
  Other Names: Oxis
  Arms: F 9.0 bid
Drug: Turbuhaler® placebo — placebo inhaled twice daily
  Arms: PBO

SUMMARY:
The purpose of this study is to show the efficacy and safety of formoterol for the maintenance treatment of patients with COPD compared with placebo in patients in Japan and in European countries during 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged above 40 with a clinical diagnosis of COPD and current COPD symptoms
* Current or previous smoker with a smoking history of 10 or more pack years
* Lung function parameters: FEV1/FVC < 70%, post-bronchodilator and post-bronchodilator FEV1 < 80% of predicted normal value

Exclusion Criteria:

* History and/or current clinical diagnosis of asthma or atopic diseases such as allergic rhinitis
* Use of inhaled glucocorticosteroids within 4 weeks prior to Visit 2
* Any relevant cardiovascular disorder as judged by the investigator or any current respiratory tract disorder other than COPD.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Goran Carlsson, MD, Study Director — AstraZeneca R&D Lund, Sweden; Miron A Bogdan, MD, Principal Investigator — Clinica Medic Or, Calea
Locations (47):
- Bulgaria (8):
  - Research Site, Gabrovo
  - Research Site, Lovech
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Troyan Municipality
  - Research Site, Varna
- Japan (28):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Seto, Aichi-ken
  - Research Site, Noda, Chiba
  - Research Site, Touon, Ehime
  - Research Site, Yanagawa, Fukuoka
  - Research Site, Ōta, Gunma
  - Research Site, Ōwa, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Chitose, Hokkaido
  - Research Site, Obihiro, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Yabu, Hyōgo
  - Research Site, Naka-gun, Ibaraki
  - Research Site, Morioka, Iwate
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Kawasaki, Kangawa
  - Research Site, Kochi, Kochi
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Katano, Osaka
  - Research Site, Kishiwada, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Takatsuiki, Osaka
  - Research Site, Chiyoda City, Tokyo
  - Research Site, Wakayama, Wakayama
  - Research Site, Ube, Yamaguchi
- Romania (4):
  - Research Site, Deva, Hunedoara County
  - Research Site, Bucharest
  - Research Site, Constanța
  - Research Site, Iași
- Russia (3):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Ukraine (4):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kyiv

REFERENCES:
- [Derived] Bogdan MA, Aizawa H, Fukuchi Y, Mishima M, Nishimura M, Ichinose M. Efficacy and safety of inhaled formoterol 4.5 and 9 mug twice daily in Japanese and European COPD patients: phase III study results. BMC Pulm Med. 2011 Nov 15;11:51. doi: 10.1186/1471-2466-11-51. PMID 22085439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients, male or female aged ≥ 40 years with moderate to severe chronic obstructive pulmonary disease (COPD). 766 subjects enrolled; 153 excluded: 96 for incorrect enrollment, 17 for adverse events, 32 for voluntary discontinuation, 1 for non-compliance with protocol, 7 for other reasons. 613 were randomised.
Groups:
- Formoterol 4.5 Bid: Formoterol 4.5 ug bid
- Formoterol 9.0 Bid: Formoterol 9.0 ug bid
- Placebo: Placebo
Period: Overall Study
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Started | 206 (randomised patients) | 199 (randomised patients) | 208 (randomised patients)
Completed | 195 (randomised patients) | 182 (randomised patients) | 186 (randomised patients)
Not Completed | 11 | 17 | 22
Not completed — Adverse Event | 6 | 8 | 10
Not completed — Withdrawal by Subject | 4 | 6 | 11
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — COPD Exacerbation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo | Total
Number analyzed (Participants) | 206 | 199 | 208 | 613
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (9.4) | 67.2 (9.2) | 66.3 (9.7) | 66.75 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 29 | 22 | 74
  Male | 183 | 170 | 186 | 539

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1; L) 60 Minutes Post-dose
Description: FEV1 (expressed as litres [L]) is a spirometric measure of lung function. FEV1 was measured 60 minutes after administration of study drug. The results are expressed as a percentage in relation to the baseline value.
Time Frame: from baseline up to 12 weeks
Measure: Geometric Mean (Full Range); unit: percent of baseline
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 199 | 208
percent of baseline | 112.9 [75.1 to 177.0] | 113.36 [66.2 to 184.0] | 101.28 [58.3 to 189.1]

2. Secondary Outcome: Forced Vital Capacity (FVC) 60 Minutes Post-dose
Description: Forced Vital Capacity (FVC) is a spirometric measure of lung function. FVC was measured 60 minutes after administration of study drug. The results are expressed as a percentage in relation to the baseline value
Time Frame: from baseline up to 12 weeks
Measure: Geometric Mean (Full Range); unit: percent of baseline
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 199 | 208
percent of baseline | 109.73 [81.2 to 162.0] | 109.92 [83.2 to 200.9] | 102.11 [71.2 to 212.7]

3. Secondary Outcome: FEV1 Pre-dose
Description: Lung function (FEV1) was measured before administrations of the study drug (pre-dose). The results are expressed as a percentage of mean FEV1 over visists 4-6 in relation to the baseline (visit 3) value
Time Frame: baseline at week 0 and pre-dose at weeks 4, 8 and 12
Measure: Geometric Mean (Full Range); unit: percent of baseline
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 196 | 204
percent of baseline | 104.54 [73.3 to 175.0] | 104.65 [71.0 to 172.6] | 99.77 [56.5 to 183.6]

4. Secondary Outcome: FVC Pre-dose
Description: Lung function (FVC) was measured before administrations of the study drug (pre-dose). The results are expressed as a percentage of mean FEV1 over visists 4-6 in relation to the baseline (visit 3) value
Time Frame: baseline at week 0 and pre-dose at weeks 4, 8 and 12
Measure: Geometric Mean (Full Range); unit: percent of baseline
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 196 | 204
percent of baseline | 103.62 [77.7 to 149.8] | 103.36 [68.9 to 162.7] | 100.73 [70.8 to 211.9]

5. Secondary Outcome: FEV1 5 Minutes Post-dose
Description: Lung function (FEV1) was measured 5 minutes after the first dose of study drug. The results are expressed as a percentage in relation to the baseline value
Time Frame: baseline and 5 minutes anter first dose
Measure: Geometric Mean (Full Range); unit: percent of baseline
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 197 | 207
percent of baseline | 110.16 [65.6 to 156.5] | 110.24 [80.6 to 155.1] | 101.25 [79.4 to 121.6]

6. Secondary Outcome: FVC 5 Minutes Post-dose
Description: Lung function (FVC) was measured 5 minutes after the first dose of study drug, The results are expressed as a percentage in relation to the baseline value
Time Frame: baseline and 5 minutes anter first dose
Measure: Geometric Mean (Full Range); unit: percent of baseline
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 197 | 207
percent of baseline | 108.50 [89.9 to 143.2] | 108.88 [81.5 to 153.4] | 101.59 [84.3 to 124.7]

7. Secondary Outcome: Change in Peak Expiratory Flow (PEF), Morning
Description: Patients were asked to measure and record lung function (peak expiratory flow [PEF] measured in the morning). Average values over the last 10 days of the run-in period and the whole treatment period were calculated. The results are expressed as the change from the run-in period average value
Time Frame: run-in period and 12 week
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 198 | 205
L/min | 16.27 (27.90) | 18.34 (26.19) | 3.60 (27.08)

8. Secondary Outcome: Change in Peak Expiratory Flow (PEF), Evening
Description: Patients were asked to measure and record lung function (peak expiratory flow [PEF] measured in the evening). Average values over the last 10 days of the run-in period and the whole treatment period were calculated. The results are expressed as the change from the run-in period average value
Time Frame: run-in period and 12 week
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 198 | 205
L/min | 13.15 (27.52) | 15.76 (25.22) | 2.36 (26.43)

9. Secondary Outcome: Change in Night-time Awakenings Due to Symptoms
Description: Patients were asked to record the night-time awakenings due to symptoms (scored from 0-4 with 4 being the most severe). Period averages over the last 10 days of the run-in period and the whole treatment period were calculated. The results are expressed as the change from the run-in period average value
Time Frame: run-in period up to 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale per day
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 198 | 207
scores on a scale per day | -0.1318 (0.4791) | -0.1748 (0.5517) | -0.0466 (0.4900)

10. Secondary Outcome: Breathlessness
Description: Patients were asked to record breathlessness (scored from 0-4 with 4 being the most severe). Period averages over the last 10 days of the run-in period and the whole treatment period were calculated. The results are expressed as the change from the run-in period average value
Time Frame: run-in period up to 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale per day
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 198 | 207
scores on a scale per day | -0.4068 (0.6193) | -0.4531 (0.5511) | -0.2626 (0.5899)

11. Secondary Outcome: Cough
Description: Patients were asked to record cough (scored from 0-4 with 4 being the most severe). Period averages over the last 10 days of the run-in period and the whole treatment period were calculated. The results are expressed as the change from the run-in period average value
Time Frame: run-in period up to 12 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale per day
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 206 | 198 | 207
scores on a scale per day | -0.3250 (0.6424) | -0.4088 (0.6374) | -0.2016 (0.6233)

12. Secondary Outcome: Use of Reliever Medication
Description: Patients were asked to record reliever medication use. Period averages over the last 10 days of the run-in period and the whole treatment period were calculated. The results are expressed as the change from the run-in period average value
Time Frame: 12 weeks (end of run-in to last visit)
Measure: Mean (Standard Deviation); unit: medication doses per day
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 204 | 196 | 207
medication doses per day | -0.60 (1.47) | -0.97 (1.88) | -0.23 (1.25)

13. Secondary Outcome: St George's Respiratory Questionnaire (SGRQ)
Description: Patients were asked to complete the St George's Respiratory Questionnaire (SGRQ). Subscale symptom score ranges from 0 to 100% and measures the effect of respiratory symptoms, frequency, and severity on quality of life. A score of 0 indicates the best possible status. Results are expressed as the change from baseline score with a decrease in score indicating improvement.
Time Frame: 12 weeks (end of run-in to last visit)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Number analyzed (Participants) | 203 | 191 | 206
Scores on a scale | -5.46 (12.12) | -6.38 (10.77) | -2.02 (12.98)

ADVERSE EVENTS:
Arm/Group | Formoterol 4.5 Bid | Formoterol 9.0 Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 6/206 | 7/199 | 4/208
Other Adverse Events (participants affected / at risk) | 33/206 | 31/199 | 31/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Formoterol 4.5 Bid (N=206) | Formoterol 9.0 Bid (N=199) | Placebo (N=208)
Death (General disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate Caner (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemic Unconsciousness (Metabolism and nutrition disorders) | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Formoterol 4.5 Bid (N=206) | Formoterol 9.0 Bid (N=199) | Placebo (N=208)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 15
Nasopharyngitis (Infections and infestations) | 24 | 25 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less